CLINICAL TRIAL: NCT03325270
Title: Effect of Prebiotics on Iron Absorption in Women With Low Iron Stores
Acronym: Fe_GOS_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Burgerstein Vitamine (Industry)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Head of Laboratory of Human Nutrition, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Fe_GOS_1
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Iron-deficiency
Keywords: prebiotics; Galacto-oligosaccharides; Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ferrous fumarate (Experimental): labeled iron as Ferrous Fumarate
  Interventions: Dietary Supplement: labeled ferrous fumarate
- ferrous fumarate and GOS (Experimental): labeled ferrous fumarate + prebiotics
  Interventions: Dietary Supplement: labeled ferrous fumarate + prebiotics
- ferrous sulfate and GOS (Experimental): labeled ferrous sulfate + prebiotics
  Interventions: Dietary Supplement: labeled ferrous sulfate + prebiotics

INTERVENTIONS:
Dietary Supplement: labeled ferrous fumarate — labeled iron as Ferrous Fumarate
  Arms: ferrous fumarate
Dietary Supplement: labeled ferrous fumarate + prebiotics — labeled iron as Ferrous Fumarate + galacto-oligosaccharides
  Arms: ferrous fumarate and GOS
Dietary Supplement: labeled ferrous sulfate + prebiotics — labeled iron as Ferrous Sulfate + galacto-oligosaccharides
  Arms: ferrous sulfate and GOS

SUMMARY:
Rationale:

According to the WHO, iron deficiency is still the most common and widespread nutritional disorder in the world. Current iron supplements have limitations in terms of bioavailability and tolerability. Prebiotic fibers, such as galacto-oligosaccharides (GOS), selectively enhance growth of beneficial colonic bacteria. Prebiotics in general enhance the production of short-chain fatty acids (SCFAs) and thereby decrease luminal pH. Through the reduction in colonic pH, prebiotics can enhance absorption of minerals such as calcium and magnesium and they have been proposed to potentially improve iron absorption as well.

The primary objective of this study is to investigate the effect of an addition of GOS to an iron supplement on iron absorption in iron deplete, healthy, normal weight women.

DETAILED DESCRIPTION:
Iron deficiency is still the most common and widespread nutritional disorder in the world according to WHO. It does not only affect large numbers of women and children in the developing world, but also in industrialized countries. The current estimation is that 2 billion people, or around 30% of the world's population, are anemic, of which around 50% is caused by iron deficiency. In industrialized countries, ID remains a public health concern in young women, affecting 16% of females between the ages of 12-49y in the United states.

Iron supplementation has been recommended by the WHO as an approach to improve iron status in varying age and risk groups. Iron supplementation can be practical for high-risk groups such as pregnant women and has been proven effective for increasing hemoglobin levels in women. However, iron absorption from supplements is generally low and epigastric side effects reduce compliance. With the high global burden of iron deficiency and anemia, improved products which allow better absorption and reduce side effects are urgently needed.

Targeted iron supplementation in high risk groups is the preferred way to treat iron deficiency. However, the recommendation is to consume iron supplements away from food in order to increase bioavailability which often causes nausea and epigastric pain and thus reduces compliance. Taken together with food, bioavailability of most supplements is reduced by about two thirds. Thus, a lot of unabsorbed iron passes into the colon where it can increase the abundance of enteropathogens.

Prebiotic fibers, such as galacto-oligosaccharides (GOS), selectively enhance growth of beneficial colonic bacteria. GOS are enzymatically produced from lactose and are a mixture of glucose- and galactose- based di- and oligosaccharides of varying structure and seem to have an increased selectivity towards Bifidobacterium spp compared to other prebiotics. Prebiotics in general enhance the production of short-chain fatty acids (SCFAs) and thereby decrease luminal pH, which may reduce growth of enteropathogens. Through the reduction in colonic pH, prebiotics can enhance absorption of minerals such as calcium and magnesium and they have been proposed to potentially improve iron absorption, by reducing ferric to ferrous iron in the colon. Even though colonic absorption is minimal compared to absorption in the duodenum in healthy humans, it may become more important in iron deficiency or anemia as demonstrated in animal studies.

The primary objective of this study is to investigate the effect of an addition of GOS to an iron supplement on iron absorption in iron deplete, healthy, normal weight women.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* SF levels <20 µg/L
* Normal body Mass Index (18.5-24.9 kg/m2)
* Body weight <70 kg
* Signed informed consent

Exclusion Criteria:

* Severe anaemia (Hb < 80 g/L)
* Elevated CRP >10.0 mg/L
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole studies (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration, including pre- and-or probiotics supplements (excluding foods and beverages with life cultures such as yoghurt, raw milk cheese and kombucha)
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Difficulties with blood sampling
* Use of antibiotics over the past month
* Known hypersensitivity to iron supplements in the given amount, GOS, or lactose
* Women who are pregnant or breast feeding
* Women who intend become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse -
* Smokers (> 1 cigarette per week)
* Inability to follow the procedures of the study, e.g. due to language problems, self-reported psychological disorders, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are being studied
Enrollment: 46 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
fractional iron absorption | 2 months
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of several isotopically labelled iron supplements (days 0, 2 16, 18, 20, 37, 39, 41).Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeroense FMD, Michel L, Zeder C, Herter-Aeberli I, Zimmermann MB. Consumption of Galacto-Oligosaccharides Increases Iron Absorption from Ferrous Fumarate: A Stable Iron Isotope Study in Iron-Depleted Young Women. J Nutr. 2019 May 1;149(5):738-746. doi: 10.1093/jn/nxy327. PMID 31004135